CLINICAL TRIAL: NCT03204812
Title: A Pilot Trial to Explore the Link Between Immunological Changes, Efficacy, Safety, and Tolerability of Durvalumab (MEDI4736) Plus Tremelimumab in Chemotherapy-Naïve Men With Metastatic Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Durvalumab and Tremelimumab in Treating Chemotherapy Naive Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0769; NCI-2018-01135 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0769 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-10

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Prostate Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tremelimumab, durvalumab) (Experimental): Patients receive tremelimumab IV over 60 minutes and durvalumab IV over 60 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles for tremelimumab and up to 13 cycles for durvalumab in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This phase II trial studies the safety, tolerability and how well durvalumab and tremelimumab work in treating participants with castration-resistant prostate cancer who have not received chemotherapy (chemotherapy naïve) and has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as durvalumab and tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of durvalumab plus tremelimumab in patients with metastatic castration-resistant prostate cancer.

SECONDARY OBJECTIVES:

I. To assess the efficacy of durvalumab plus tremelimumab in patients with metastatic castration-resistant prostate cancer. II. To explore immunological changes in peripheral blood and tissue (e.g. peripheral blood cluster of differentiation [CD] 4+ [Inducible COStimulator (ICOS)]+ T cells, CD3 expression in tissue) in response to durvalumab plus tremelimumab in patients with metastatic castration-resistant prostate cancer.

OUTLINE:

Patients receive tremelimumab intravenously (IV) over 60 minutes and durvalumab IV over 60 minutes on day 1. Treatment repeats every 28 days for up to 4 cycles for tremelimumab and up to 13 cycles for durvalumab in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 60, and 90 days, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of >= 52 weeks.
* Hemoglobin >= 11.0 g/dL.
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (> 1500 per mm^3).
* Platelet count >= 100 x 10^9/L (>100,000 per mm^3).
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]/alanine aminotransferase [ALT] serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal.
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Consent to MD Anderson laboratory protocol PA13-0291 and LAB02-152.
* Willing to have peripheral blood mononuclear cells and bone marrow biopsies to be collected prior to receiving the first dose of durvalumab and tremelimumab, after 2-doses and 4-doses of durvalumab and tremelimumab, after 2nd treatment administration and 4th treatment administration.
* Histologically or cytologically confirmed adenocarcinoma of the prostate.
* Evidence of metastatic disease to the bone seen on most recent bone scan, computed tomography (CT) scan and/or magnetic resonance imaging (MRI).
* Asymptomatic or minimally symptomatic patients (do not require narcotics for prostate cancer-related pain).
* Tumor progression while on hormone therapy with castrate levels serum testosterone (=< 1.7 nmol/L or 50 ng/dL) defined by prostate-specific antigen (PSA) and/or radiographic criteria according to the Prostate Cancer Working Group 3 (PCWG3). Castrate levels of testosterone must be maintained by surgical or medical means throughout the conduct of the study.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site), previous enrollment in the present study.
* Participation in another clinical study with an investigational product during the last 4 weeks.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab.
* History of another primary malignancy except for: 1) Malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence. 2) Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease. 3) Adequately treated carcinoma in situ without evidence of disease (e.g., superficial bladder cancer).
* Evidence of visceral metastasis to the liver.
* Prior use of taxane-based chemotherapy for treatment of castrate resistant prostate cancer.
* Receipt of the last dose of anti-cancer therapy (immunotherapy, endocrine therapy [e.g., abiraterone acetate, enzalutamide], targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) =< 28 days prior to the first dose of study drug. (with the exception of any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab.)
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of durvalumab or tremelimumab. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* QT interval corrected for heart rate using Fridericia's formula (QTcF) >= 470 ms. Any clinically significant abnormalities detected, require triplicate electrocardiogram (ECG) results and a mean QT interval corrected for heart rate using Fridericia's formula (QTcF) >= 470 ms calculated from 3 electrocardiograms (ECGs).
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of: intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid or steroids as pre-medication for hypersensitivity reactions (e.g. CT scan premedication).
* Any unresolved toxicity (Common Terminology Criteria for Adverse Events [CTCAE] grade >= 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy).
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia;
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement;
  * Any chronic skin condition that does not require systemic therapy;
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician;
  * Patients with celiac disease controlled by diet alone.
  * Subjects with history of diverticulitis may be included only after consultation and approval of the study physician.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of hypersensitivity to the combination of durvalumab and tremelimumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diathesis including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Known history of positive test for hepatitis B virus (HBV) using HBV surface antigen (HBV sAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection.
* History of leptomeningeal carcinomatosis.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 28 days prior to study treatment start. Patients with suspected brain metastases at screening should have a CT/MRI of the brain prior to study entry.
* Subjects with uncontrolled seizures.
* Male patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.
* A malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 years, or has a >= 30% probability of recurrence within 24 months (except for non-melanoma skin cancer or Ta urothelial carcinomas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumit K Subudhi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Subudhi SK, Siddiqui BA, Aparicio AM, Yadav SS, Basu S, Chen H, Jindal S, Tidwell RSS, Varma A, Logothetis CJ, Allison JP, Corn PG, Sharma P. Combined CTLA-4 and PD-L1 blockade in patients with chemotherapy-naive metastatic castration-resistant prostate cancer is associated with increased myeloid and neutrophil immune subsets in the bone microenvironment. J Immunother Cancer. 2021 Oct;9(10):e002919. doi: 10.1136/jitc-2021-002919. PMID 34663638
- See also: The University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: July 2017- April 2019
Pre-assignment Details: 31 participants consented, 5 participants were inevaluable.
Period: Overall Study
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Started | 26
Completed | 23
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 67.5 [48 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Toxicity will be monitored in all patients who receive at least one dose of tremelimumab, even if the patient is not evaluable for the biomarker or efficacy endpoint. Will be assessed per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03.
Time Frame: from date of the first treatment, up to 43.6 months
Population: One patient received only one dose of combination therapy and was excluded from efficacy analysis.
Measure: Number; unit: adverse events
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 25
adverse events
  Adverse Events | 236
  Serious Adverse Events | 14

2. Secondary Outcome: Prostate-specific Antigen (PSA) Progression Free Survival (PFS)
Description: PSA PFS is defined as per Prostate Cancer Working Group 3 (PCWG3) criteria: time from start of therapy to first PSA increase of 25% and ≥2 ng/mL above the nadir, and which is confirmed by a second value ≥3 weeks later. PSA PFS were calculated from the first day of treatment and summarized by Kaplan-Meier methods.
Time Frame: from the first day of treatment, up to 43.6 months
Population: One patient received only one dose of combination therapy and was excluded from efficacy analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 25
months | 0.9 [0.9 to 1.8]

3. Secondary Outcome: Radiographic Progressive Free Survival (rPFS)
Description: rPFS is measured from first dose to date of disease progression on CT and/or bone scan or death from any cause, whichever occurs first. Radiographic PFS will start at the first day of treatment and will be summarized by Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1),as a 20% increase in the sum of the longest diameter of target lesions, or ameasurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: from first day of treatment, up to 43.6 months
Population: One patient received only one dose of combination therapy and was excluded from efficacy analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 25
months | 3.7 [1.9 to 5.7]

4. Secondary Outcome: Number of Participants With PSA Decline of ≥50% From Start of Therapy
Description: PSA decline will start at the first day of treatment and will be summarized by Kaplan-Meier. The numeric PSA value at maximal decline will be summarized by a boxplot and as a scatter plot of maximal decline by baseline PSA. PSA is produced by normal and cancerous prostate tissue. PSA levels are often elevated in men with prostate cancer.
Time Frame: baseline, up to 43.6 months
Population: One patient received only one dose of combination therapy and was excluded from efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 25
Participants | 3

5. Secondary Outcome: Median Overall Survival
Description: Overall Survival is the time which begins at diagnosis (or at the start of treatment) and up to the time of death.
Time Frame: from start of treatment, up to 43.6 months
Population: One patient received only one dose of combination therapy and was excluded from efficacy analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Tremelimumab, Durvalumab)
Number analyzed (Participants) | 25
months | 28.1 [14.5 to 37.3]

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of medication, up to 43.6 months
Arm/Group | Treatment (Tremelimumab, Durvalumab)
All-Cause Mortality (participants affected / at risk) | 14/26
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tremelimumab, Durvalumab) (N=26)
Colitis (Gastrointestinal disorders) | 2 (3)
Diabetes type 1 (Endocrine disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Lipase increased (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Spinal Cord Compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tremelimumab, Durvalumab) (N=26)
Alanine aminotransferase increased (Investigations) | 5 (7)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 10 (17)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (3)
Blurred vision (Eye disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Investigations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 8 (13)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Increased cortisol (Endocrine disorders) | 5 (6)
Decreased cortisol (Endocrine disorders) | 4 (5)
Hypophysitis (Endocrine disorders) | 2 (2)
Decreased ACTH (Endocrine disorders) | 2 (2)
Increased non-fasting blood glucose (Endocrine disorders) | 2 (2)
Diabetes Type 1 (Endocrine disorders) | 1 (1)
T4 decrease (Endocrine disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
GGT increased (Investigations) | 2 (4)
Headache (Nervous system disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased sedimentation rate (Investigations) | 1 (1)
Increased sedimentation rate (Investigations) | 4 (4)
Increase CK (Investigations) | 1 (1)
Increase Aldolase (Investigations) | 1 (1)
Alkaline phosphate increase (Investigations) | 1 (1)
ACTH Elevated (Investigations) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lipase increased (Investigations) | 6 (14)
Lymphocyte count decreased (Investigations) | 3 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (14)
Respiratory, thoracic and mediastinal disorders - Other, pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 6 (11)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT03204812/Prot_SAP_000.pdf